CLINICAL TRIAL: NCT05074992
Title: A Phase II Trial of Neoadjuvant Therapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Trial of Neoadjuvant Therapy in Patients With Newly Diagnosed Glioblastoma
Acronym: NeAT Glio
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Support withdrawn from drug company supplying IMP
Sponsor: University College, London (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/134643
Record Dates: First submitted 2021-06-25; First posted 2021-10-12 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
Keywords: Newly Diagnosed
MeSH Terms: conditions — Glioblastoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ipilimumab (Experimental): 3mg/kg Ipilimumab IV infusion (day 1) given as a 21 day cycle for 2 cycles.
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab is a monoclonal antibody medication that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system.

SUMMARY:
The NeAT Glio trial will evaluate whether the addition of ipilimumab prior to the current standard treatment of surgery and chemoradiotherapy will improve survival in patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
This is a phase II trial to evaluate whether the addition of ipilimumab prior to the current standard treatment of surgery and chemoradiotherapy will improve survival in patients with newly diagnosed glioblastoma.

The trial will recruit 43 patients over 1 year.

Trial Subjects (patients) with newly diagnosed de-novo glioblastoma who are deemed eligible for the trial will be recruited to the study to receive neoadjuvant ipilimumab. Patients will receive 2 cycles of ipilimumab, administered intravenously at a dose of 3mg/kg on day 1 of each 21 day cycle.

Prior to trial entry the patient's treating multidisciplinary team (MDT) consisting of oncologists, radiologists and surgeons must agree that the patient is a suitable candidate for ipilimumab prior to surgery and that surgery may be delayed beyond usual standard of care timelines.

Patients will be assessed on a weekly basis, and disease assessments (including MRI scans) will be performed after each cycle of ipilimumab. Patient responses and associated MRI scans will be reviewed by the MDT to determine that it is safe for the patient to continue with trial treatment. On completion of trial treatment patients will have a further disease assessment (including MRI scan) which will be reviewed with the MDT before continuing to standard of care treatment of debulking surgery and chemoradiation.

Patients demonstrating clinical or radiological deterioration (as determined by the MDT or the principal investigator) at any point, either before starting or whilst receiving ipilimumab, will stop trial treatment and proceed to debulking surgery and chemoradiotherapy as per local policies.

Patients will be followed up every 3 months for 2 years and then annually thereafter.

End of trial will be declared when the final data item for the final patient is received i.e. when the final patient completes their 2 year follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, newly diagnosed de-novo supratentorial glioblastoma (including gliosarcoma)
2. Age ≥18 years
3. Tumour deemed appropriate for surgical debulking
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. Clinically fit for, and appropriate to receive, neoadjuvant ipilimumab followed by standard of care treatment, based on investigator and MDT judgement
6. Adequate organ and bone marrow function: Hb ≥9 g/dL, neutrophils ≥1.0 x 10 9/L, platelets ≥100 x 10 9/L and lymphocyte count ≥1.0 x 10 9/L
7. Adequate renal function: < 1.5 x ULN or a creatinine clearance of ≥ 50mL/min calculated by Cockroft-Gault equation
8. Adequate liver function, including:

   1. Bilirubin ≤ 1.5 x ULN (except for patients with known Gilbert's Syndrome who may have total bilirubin ≤ 3 x ULN)
   2. Aspartate or alanine transferase (AST or ALT) ≤ 2.5 x ULN
9. Life expectancy of greater than 12 weeks
10. Willing to comply with the contraceptive requirements of the trial
11. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
12. Willing to donate tumour material and serial blood samples
13. Written informed consent

Exclusion Criteria:

1. Diagnosis of Multifocal glioblastoma (Multicentric glioblastoma permitted)
2. Prior resection of glioblastoma leaving inadequate tissue for post investigational treatment resection
3. Secondary glioblastoma (i.e. previous histological or radiological diagnosis of lower grade glioma)
4. Known extracranial metastatic or leptomeningeal disease
5. Prior treatment for glioblastoma other than a limited resection or biopsy
6. Dexamethasone dose >3mg daily (or equivalent) at the time of starting study treatment
7. Antibiotics within 30 days of starting study treatment
8. Intratumoural or peritumoural haemorrhage deemed significant by the treating physician
9. Active autoimmune disease apart from:

   1. Skin conditions such as psoriasis, vitiligo or alopecia not requiring systemic treatment
   2. Type 1 diabetes or thyroid disease, controlled on medication
10. Any evidence of severe or uncontrolled diseases (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
11. Known hypersensitivity to ipilimumab or any of its excipients
12. Past medical history of interstitial lung disease, idiopathic pulmonary fibrosis, drug-induced interstitial disease which required steroid treatment or any evidence of clinically active interstitial lung disease
13. Any condition requiring systemic treatment with corticosteroids (>10mg prednisolone daily or equivalent) or other immunosuppressive medications within 14 days of starting study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10mg daily prednisolone or equivalent are permitted in the absence of active autoimmune disease
14. Treatment with any other investigational agent within 28 days prior to starting study treatment
15. History of previous cancer within 5 years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions
16. Positive serology for Hepatitis B defined as a positive test for HepB surface antigen (HBsAg). Note: patients who are HepB core antibody (HBcAb) positive will only be eligible for the study if the HepB virus deoxyribonucleic acid (DNA) test is negative and patients are willing to undergo monthly monitoring for Hepatitis B virus reactivation
17. Positive serology for Hepatitis C defined as a positive test for Hepatitis C virus antibody
18. Diagnosis of prior immunodeficiency or organ-transplant requiring immunosuppressive therapy or known HIV or acquired immunodeficiency syndrome (AIDS)-related illness
19. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
20. Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Survival rate at 24 months | 24 months after diagnostic biopsy
  Number of patients alive at 24 months

SECONDARY OUTCOMES:
Survival rate at 12 months | 12 months after diagnostic biopsy
  Number of patients alive at 12 months
Time to treatment failure | 1st diagnostic biopsy to early treatment discontinuation, progression, starting further treatment or death up to 24 months
  Time from 1st diagnostic biopsy to early treatment discontinuation, progression, starting further treatment or death
Best Overall Objective Response Rate | After ipilimumab treatment through to study completion, an average of 36 months
  Number of patients who experienced a Complete Response (CR), Partial Response (PR), Minor Response (MR) or Stable Disease (SD)
Treatment emergent adverse events | From start of treatment until 3 months post administration of ipilimumab
  Adverse events being report during and after treatment, coded using CTCAE v5.0
Treatment Compliance | From start of treatment until treatment discontinuation, an average of 2 months
  Median time on treatment for all patients
Changes in Performance Status | From screening through to study completion, an average of 3 years
  Percentages of World Health Organisation (WHO) performance status will be measured
Surgical complications | From surgery through to study completion, an average of 3 years
  Each type of surgical complication and worst severity grade will be reported, coded using CTCAE v5.0 for patients that undergo surgery
Resection rate | At the time of surgery
  Number of patients who had no surgery, achieved subtotal resection and achieved gross total resection

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mulholland, Principal Investigator — University College London Hospitals
Locations (4):
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Queen's Hospital, Romford

IPD SHARING:
Plan to Share IPD: No